CLINICAL TRIAL: NCT04098926
Title: Evaluation of Dose Integrated Accelerated Irradiation in Older Women (≥ 70 Year) With Early and Loco-regionally Advanced Stages of Breast Cancer
Brief Title: Highly Accelerated Dose-Integrated Radiotherapy in 5 Fractions in Breast Cancer
Acronym: HAI-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2014/1167
Record Dates: First submitted 2015-06-02; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2015-06

CONDITIONS: Breast Cancer; Radiotherapy
Keywords: Older women; Accelerated radiotherapy; Dose-integrated radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accelerated dose-integrated radiotherapy - pN0 (Experimental): Lymph node negative breast cancer
  Interventions: Radiation: Dose-integrated accelerated EBRT in pN0 breast cancer
- Accelerated dose-integrated radiotherapy - pN1 (Experimental): Lymph node positive breast cancer
  Interventions: Radiation: Dose-integrated accelerated EBRT in pN+ breast cancer

INTERVENTIONS:
Radiation: Dose-integrated accelerated EBRT in pN0 breast cancer — WBI: 5 x 5.7Gy Thoracic wall: 5 x 5.7Gy R0 boost: 5 x 6.5Gy R1 boost: 5 x 6.9Gy
  Arms: Accelerated dose-integrated radiotherapy - pN0
Radiation: Dose-integrated accelerated EBRT in pN+ breast cancer — WBI: 5 x 5.7Gy Thoracic wall: 5 x 5.7Gy R0 boost: 5 x 6.5Gy R1 boost: 5 x 6.9Gy Lymph node region: 5 x 5.4Gy
  Arms: Accelerated dose-integrated radiotherapy - pN1

SUMMARY:
Adjuvant radiotherapy in breast cancer improves local control, also in the elderly. Hormonal therapy in hormone sensitive tumors improves results but can not substitute radiotherapy. Improved local control leads to less breast cancer related morbidity and mortality, also in an older population (Schonberg, JCO, 2011).

Unfortunately, in older patients with lower life expectancy, adjuvant radiotherapy is often omitted. Following reasons are invoked:

* frailty of the patient
* fear for toxicity
* impaired mobility, rendering transportation and positioning more difficult
* dependency for transportation to and from the radiotherapy departement
* negative cost effectiveness ratio, due to high cost (especially for complex techniques and long schedules) and lower benefit (lower life expectancy)

Hypofractionation is feasible without increased toxicity, and combines better local control with patient comfort and lower costs. Further lowering the number of fractions (from 15-21 to 5) will further improve patient comfort, but is challenging when different doses are needed in the same target volume. This problem is addressed using advanced techniques permitting dose-integration.

In the elder with cancer, several unrecognized geriatric problems, including depression and cognitive impairment, can be detected by CGA . Some problems do interact with cancer treatment. In this study screening and assessment is provided to support patients and to develop an inventory of radiotherapy obstacles.

Our study includes breast cancer patients, ≥70 years old, referred for adjuvant radiotherapy after surgical treatment. A schedule of 5 fractions is offered, encompassing different targets of treatment.

DETAILED DESCRIPTION:
Adjuvant radiotherapy in breast cancer improves local control and overall survival, also in the elderly. Hormonal therapy in hormone sensitive tumors improves results but can not substitute radiotherapy (EBCTCG, Lancet, 2011). Improved local control, leads to less breast cancer related morbidity and mortality, also in an older population (Schonberg, JCO, 2011).

Unfortunately, in older patients with lower life expectancy, adjuvant radiotherapy is often perceived as too cumbersome. As a consequence, patients who could have benefit from breast conserving therapy are referred for mastectomy. Even when breast-conserving surgery is chosen, adjuvant radiotherapy is sometimes omitted in frail patients over 70 years fearing the burden of daily transportation to the radiation department. However, omitting radiotherapy results in a higher risk of loco-regional recurrence. It has been shown that older patients have a worse prognosis due to suboptimal treatment, especially in locally advanced breast cancer (Schonberg, JCO, 2011).

Following reasons are invoked by the patients or the care-givers:

* frailty of the patient
* fear for (mostly acute) toxicity
* impaired mobility, rendering transportation and positioning more difficult
* dependency on third parties (family, services) for transportation to and from the radiotherapy departement
* negative cost effectiveness ratio, due to high cost (especially for complex techniques and long schedules) and lower benefit (lower life expectancy)

Hypofractionation and acceleration are proven to be feasible in recent trials (cf. Start Trial, Fast Trial).

Based on these data and in order to overcome above mentioned obstacles for radiotherapy in breast cancer, we start a study with accelerated radiotherapy in women above 70 years old.

As we are experienced in advanced techniques as IMRT, VMAT, simultaneous dose-integration and IGRT, we will use simultaneous dose integrated protocols to permit inclusion of early as well as locally advanced breast cancer.

Integration of doses within one global volume encompasses several advantages:

* number of fractions can be maintained, regardless of the indication
* imprevisible high doses due to overlap of adjacent fields in tangential techniques is avoided
* high dose volume is more adequately limited to the actual region of high risk, as dose difference is smaller.

In order to evaluate the impact of accelerated radiotherapy on the well being of the patient and on the treatment cost, quality of life (QoL) will be measured and a cost-analysis will be performed.

Methodology of research At the radiotherapy intake consultation, patients with age ≥70 years are extensively informed on the advantages and the possible risks of accelerated irradiation. A written documentation of the study is provided to permit consultation of family and general practitioner before consent for participation. Until 1 week before the start of radiotherapy, patients can decide wether or not to participate in this study without impact on the starting day. Inclusion is performed after signing the informed consent.

The aim is to include 70 patients aged ≥ 70 years, who, after signing the informed consent, will be treated with the accelerated schemes over 10 days (5 sessions, every other day). Following doses are prescribed

* Breast: 5x5,7Gy
* R0 boost: 5x6.5Gy
* R1 boost: 5x6.9Gy
* Thoracic wall: 5x5.7Gy
* Lymph nodes: 5x5.4Gy --> these doses are simultaneously integrated, and regions are prescribed according to our standard protocol .

Positioning of the patient depends on technical possibilities and patient rigidity:

* for breast irradiation without lymph nodes, prone positioning is preferred if feasible, if not the patient is positioned in supine
* for thoracic irradiation with or without lymph node irradiation, patient is always installed in supine position
* for breast + lymph node irradiation, patients are installed in supine position.

End points of our study are acute and chronic toxicity, loco-regional control and QoL.

The study is divided in two different strata (first group without lymph node irradiation, second group with lymph node irradiation) for following reasons:

1. these groups represent different outcomes with lymph node invasion having a negative impact on morbidity, loco-regional control and overall survival
2. a higher frequency of acute moist desquamation might occur in the second group (lymph nodes included) as compared to the first group, due to a larger target volume.
3. the brachial plexus is a special concern, as it lies close or even within the target volume. Therefore we will monitor closely the effects on the brachial plexus for the second group. Nevertheless, as the total dose is lower than with normo-fractionation, the risk for brachial neuropathy is maximally reduced.

Groups

* 40 patients in group 1: irradiation of breast/thoracic wall with or without integrated boost without lymph node irradiation
* 30 patients in group 2: irradiation of breast/thoracic wall with or without integrated boost and with lymph node region irradiation

An application for funding to perform geriatric assessment is introduced. In the elder with cancer, several unrecognized geriatric problems, including depression and cognitive impairment, can be detected bij CGA . Some of these problems even interact with cancer treatment. In this study screening and assessment is provided to develop an inventory of obstacles for undergoing radiotherapy.

When screening scores positive (G8 score ≤ 14/17) geriatric assessment will be performed to evaluate the problems and needs of the patient. Patients will be referred for appropriate treatment and support. As described by Schönberg, treatment in early stage breast cancer might even lead to improved morbidity and mortality when compared to a non-cancer population, due to the 'healthy user' effect, detecting otherwise unrevealed problems. In the scope of this study, this effect can not be evaluated.

Power analysis To estimate the number of patients needed, we applied the Wilson score confidence interval test for binomial proportion, which is a 2-sided exact method for power analysis, using "SAS Power and Sample Size".

Group 1:

To achieve a conditional probability of 87% with an alpha-error of 0,1, a number of 35 patients would be needed. To compensate for drop-outs, we include 40 patients in this study-arm.

Group 2 To achieve a conditional probability of >95% with an alpha-error of 0,1, a number of 25 patients would be needed. To compensate for drop-outs, we include 30 patients in this study-arm.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years old
* AND breast conserving surgery or mastectomy for breast carcinoma
* AND multidisciplinary decision of adjuvant irradiation
* AND absence of distant metastases
* AND informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* Bilateral breast irradiation
* In case of mastectomy: positive resection margin, needing boost
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study
* History of previous radiation treatment to the same region

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Breast retraction (LENTSOMA) | 6 weeks post-radiotherapy
  Breast Cancer Conservative treatment.core (BCCT.core) objective measurement

SECONDARY OUTCOMES:
Acute toxicity: number of patients with clinical relevant dermatitis (CTCAE v. 4.0) | 1-8 weeks
  Assessment of grade of dermatitis
Acute toxicity: number of patients with moist desquamation (CTCAE v. 4.0 (grade 3) | 1-8 weeks
Acute toxicity: number of patients with pain (CTCAE v. 4.0) | 1-8 weeks
  Grade 1: mild; Grade 2: moderate, limiting activity of daily living (ADL); grade 3: severe, limiting ADL
Acute toxicity: number of patients with pruritus (CTCAE v. 4.0) | 1-8 weeks
  Grade 1: mild, localized topical intervention; Grade 2: intense, oral intervention, skin changes
Acute toxicity: number of patients with fatigue (MFI-20) | 1-8 weeks
  Questionnaire (20 questions)
Chronic toxicity: measurement of patient satisfaction with breast esthetic outcome: BREAST-Q questionnaire | Before radiotherapy and after 2 and 5 years
  BREAST-Q questionnaire: Patient reported outcome, evaluating satisfaction with esthetic outcome.
Chronic toxicity: prevalence of fibrosis | 2 and 5 years
  LENT Soma: fibrosis (score 0-3)
Chronic toxicity: prevalence of pain | 2 and 5 years
  LENT Soma: score 0-4
Chronic toxicity: prevalence of telangiectasia | 2 and 5 years
  LENT Soma: Score 0-3
Chronic toxicity: prevalence of lymphedema | 2 and 5 years
  LENT Soma: score 0-4
Chronic toxicity: prevalence of fatigue (MFI-20) | 2 and 5 years
  Questionnaire (20 questions)
Chronic toxicity - prevalence of radiation induced brachial plexopathy (RIBP) (standardized screening questionnaire), confirmed by electromyogram (EMG) | 2 and 5 years
  If a screening reveals unilateral pain, loss of function or muscular atrophy in the ipsilateral arm, an EMG will be performed to confirm/exclude RIBP
Loco-regional tumor control | 2 and 5 years
  Ipsilateral or regional breast recurrence
Distant tumor control | 2 and 5 years
  Distant metastases free survival
Breast cancer specific survival | 2 and 5 years
  Number of patients alive and without breast cancer recurrence at 2 and 5 years after adjuvant radiotherapy
Overall survival | 2 and 5 years
  Number of patients alive, 2 and 5 years after adjuvant radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital - Radiotherapy Department, Ghent, Belgium